CLINICAL TRIAL: NCT04057768
Title: Clinical Evaluation of Fractional Radiofrequency for the Treatment and Reduction of Acne Scars and Wrinkles
Brief Title: Fractional Radiofrequency for the Treatment and Reduction of Acne Scars and Wrinkles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VI0919
Record Dates: First submitted 2019-08-13; First posted 2019-08-15 (Actual); Results first posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Acne Scars - Mixed Atrophic and Hypertrophic; Wrinkle
Keywords: acne scars; wrinkles; rhytids; fractional RF
MeSH Terms: conditions — Hypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intervention (Other): Device: Venus Viva
  Interventions: Device: Venus Viva

INTERVENTIONS:
Device: Venus Viva — The Venus Viva™ fractional RF device has been shown in clinical studies to improve various skin conditions related to aging and alter collagen structures such as wrinkles, rhytids and scars.

SUMMARY:
The objective of this clinical study is to evaluate the efficacy of fractional RF for the treatment and reduction of acne scarring or facial wrinkles.

DETAILED DESCRIPTION:
Prospective, single centre, evaluator-blind, split face study of the efficacy of fractional radiofrequency (RF) for the treatment and reduction of acne scarring and facial wrinkles. The study will evaluate the progress of 15 subjects requesting treatment of scarring or facial wrinkles. The study will involve three treatments on both sides of the face with 3-5 week intervals between each treatment. Subjects will be followed at 6 and 12 weeks after their last treatment. Analysis will be performed on all subjects who receive at least one treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, male or female subjects over 21 years of age who are seeking treatment and reduction of their acne scarring or wrinkles.
2. Able to read, understand and voluntarily provide written Informed Consent.
3. Able and willing to comply with the treatment/follow-up schedule and requirements.
4. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment and for the duration of the study and have a negative Urine Pregnancy test at baseline.

Exclusion Criteria:

1. Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body (e.g. cochlear implant).
2. Subjects with any implantable metal device in the treatment area
3. Permanent implant in the treated area, such as metal plates and screws (excluding dental implants), or an injected chemical substance.
4. Current or history of any kind of cancer, or dysplastic nevi
5. Severe concurrent conditions, such as cardiac disorders.
6. Pregnancy or intending to become pregnant during the study and nursing.
7. Impaired immune system due to immunosuppressive diseases, such as AIDS and HIV, or use of immunosuppressive medications.
8. History of diseases stimulated by heat, such as recurrent herpes simplex in the treatment area; may be enrolled only following a prophylactic regime.
9. Poorly controlled endocrine disorders, such as diabetes.
10. Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
11. History of skin disorders, such as keloids, abnormal wound healing, as well as very dry and fragile skin.
12. History of bleeding coagulopathies, or use of anticoagulants (excluding daily aspirin).
13. Facial dermabrasion, facial resurfacing, or deep chemical peeling within the last three months, if face is treated.
14. Use of isotretinoin (Accutane®) or other systemic retinoids within six months prior to treatment or as per investigators discretion.
15. Any surgical procedure in the treatment area within the last six months or before complete healing.
16. Treating over tattoo or permanent makeup.
17. Excessively tanned skin from sun, tanning beds or tanning creams within the last two weeks.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2020-03-03 (Actual); Study Completion 2020-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Gronski, Study Director — Venus Concept
Locations (1):
- Laser and Skin Surgery Center of Northern California, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Venus Viva™ Device: Venus Viva™ Device: The Venus Viva™ fractional RF device has been shown in clinical studies to improve various skin conditions related to aging and alter collagen structures such as wrinkles, rhytids and scars.
Period: Overall Study
Arm/Group | Venus Viva™ Device
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Overall Wrinkle Improvement Assessed by the Fitzpatrick Wrinkle and Elastosis Scale (FWES) at 12 Weeks Post-Final Treatment
Description: Evaluate the efficacy of overall facial wrinkles improvement assessed live by the Investigator and a subject assessment of facial appearance including the Fitzpatrick Wrinkle and Elastosis Scale (FWES).
  The FWES is a 9 point scale.
  Three independent evaluators evaluated before and after photographs and graded them for change.
  Possible responses were: a score of 1 - 3 (Mild) indicates fine texture changes with subtly accentuated skin lines, a score of 4 - 6 (Moderate) indicates distinct papular elastosis ([indvidual papules with yellow translucency under direct lighting] and dyschromia and a score of 7 - 9 (Severe) indicates multipapular and confluent elastosis [thickened yellow and pallid] approaching or consistent with cutis rhomboidalis. A lower class and a lower score means a better outcome.
Time Frame: 12 Weeks Post-Final Treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
units on a scale
  Baseline | 5.97 (0.20)
  12-weeks | 5.78 (0.22)

2. Primary Outcome: Overall Acne Scar Improvement Assessed by the Global Aesthetic Improvement Scale (GAIS) at 12 Weeks Post-Final Treatment
Description: Evaluate the efficacy of overall facial acne scar improvement assessed live by the Investigator and a subject assessment of facial appearance including the Global Aesthetic Improvement Scale (GAIS).
  The Global Aesthetic Improvement Scale is a seven-grade subjective test.
  Three independent evaluators evaluated before and after photographs and graded them for change.
  Possible responses were (3) Very Much Improved, (2) Much Improved, (1) Improved, (0) No Change, (-1) Worse, (-2) Much Worse, and (-3) Very Much Worse. For reporting of outcomes, the higher the GAIS value, the greater the improvement (Range -3 to 3).
Time Frame: 12 Weeks Post-Final Treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
units on a scale | 0.4 (0.1)

3. Secondary Outcome: Subject Satisfaction
Description: Subjects' assessment of satisfaction with the treatment using a 5 point Subject Satisfaction Scale at 6 Weeks and 12 weeks post-treatment.
  The Subject Satisfaction Scale is a five-grade subjective test.
  Participant were asked their satisfaction level post treatment.
  Possible responses were (4) Very Satisfied, (3) Satisfied, (2) Having No Opinion, (1) Unsatisfied, and (0) Very Unsatisfied.
Time Frame: 6 and 12 Weeks Post- Final Treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
units on a scale
  6-weeks | 3.22 (0.22)
  12-weeks | 3.20 (0.25)

4. Secondary Outcome: Subject Scale - Wong Baker FACES Pain Scale
Description: Subject's assessment of discomfort and pain after treatments as measured by a 10 point Wong-Baker FACES Pain Scale
  The Wong-Baker FACES pain scoring system is a subject-reported instrument using a scale of 0 (no pain) to 10 (most pain).
  Possible responses, 9 to 10 shows Hurts Worst, 7 to 8 shows Hurts Whole Lot, 5 to 6 shows Hurts Even More, 3 to 4 shows Hurts Little More, 1 to 2 shows Hurts Little Bit, 0 shows No Hurt.
Time Frame: 12 Weeks Post-Final Treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
units on a scale | 3.93 (0.39)

5. Secondary Outcome: Subject Scale - 5 Point Scale for Treatment Tolerability
Description: Subject's assessment of treatment tolerability as measured by a 5 point scale.
  Participant were asked their tolerability level post treatment.
  Possible scores were; (4) Very Tolerable, (3) Tolerable, (2) Having No Opinion, (1) Intolerable, and (0) Very Intolerable.
Time Frame: 8 Weeks Post-Final Treatment
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 10
units on a scale | 3.10 (0.10)

6. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events
Description: Subjects experiencing a treatment-related adverse event (AE) by 12 weeks post-treatment.
  A treatment-related adverse event was any untoward medical occurrence attributed to the device in a participant who received treatment. Relatedness to the device was assessed by the investigator.
Time Frame: Up to 12 Weeks Post-Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-19): https://cdn.clinicaltrials.gov/large-docs/68/NCT04057768/Prot_SAP_000.pdf